CLINICAL TRIAL: NCT01226979
Title: Phase II Study of High-Dose-Rate Endorectal Brachytherapy (HDRBT) in the Treatment of Locally Advanced Low Rectal Cancer
Brief Title: Study of High-Dose-Rate Endorectal Brachytherapy (HDRBT) in the Treatment of Locally Advanced Low Rectal Cancer
Acronym: HDRBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0977; NA_00029263 (Other: JHMIRB)
Record Dates: First submitted 2010-09-21; First posted 2010-10-22 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; high dose endorectal brachytherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: High-Dose-Rate Endorectal Brachytherapy (HDRBT)
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HDRBT (High Dose Rectal Brachytherapy) (Experimental): Radiation: High-dose endorectal brachytherapy The investigational tool being evaluated is high-dose endorectal brachytherapy (HDRBT) which is an FDA approved method to administer endoluminal radiation for low rectal cancer. A daily dose of 6.5 Gy over four consecutive days
  Interventions: Radiation: High-dose endorectal brachytherapy (HDRBT)

INTERVENTIONS:
Radiation: High-dose endorectal brachytherapy (HDRBT) — The investigational tool being evaluated is high-dose endorectal brachytherapy (HDRBT) which is an FDA approved method to administer endoluminal radiation for low rectal cancer.
  Other Names: HDRBT

SUMMARY:
This research is being done to see how effective high-dose rate endorectal brachytherapy (HDRBT) is in treating cancer of the lowest part of the bowel (rectum). In this study we want to try to decrease side effects and shorten the course of radiation treatment for patients with cancer of their rectum by using a high-dose rate endorectal brachytherapy (HDRBT). This is a different form of radiation than what is normally given (CRT). With HDRBT, the radiation is given through an applicator placed into the bowel next to the tumor. The radiation is directed at the tumor and a small area around it.

DETAILED DESCRIPTION:
This study is a pilot study open to patients with clinical stage T2N1 or T3N0-1 resectable rectal cancer. The investigational tool being evaluated is high-dose endorectal brachytherapy (HDRBT) which is an FDA approved method to administer endoluminal radiation for low rectal cancer. This study assumes that the rate of pathological response to HDRBT will be similar to historical controls (conventional neoadjuvant chemoradiation). All patients will receive postoperative standard 5-fluorouracil (FU) based chemotherapy (at the discretion of the medical oncologist). The clinical response will be assessed with endoscopic/ultrasound, pelvic MRI and fluorodeoxyglucose (FDG)-positron emission tomography (PET)/CT. In addition, tissue and serum will be collected to evaluate for biological predictors of response to therapy. The endpoints of this study include adverse events (gastrointestinal toxicity), quality of life as measured by the quality of life questionnaire (QLQ)-C30, and tumor regression/response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed adenocarcinoma of the rectum
* Able to undergo local staging of the rectal tumor performed by MRI and/or endoscopic ultrasonography (EUS) demonstrating a T2N1 or T3N0-1 tumor
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Participants are willing to undergo initial therapy and if needed subsequent therapy prior to resection at Johns Hopkins Medical Institutions
* English as a primary language in order to complete the quality of life questionnaires

Exclusion Criteria:

* Patients with tumors >12 cm from the anal verge.
* Near obstructing or bulky tumors which will not allow application of the endorectal probe
* Patients with distant metastatic disease
* Any pelvic lymph nodes outside of the mesorectum (iliac or inguinal)
* Prior history of radiation therapy to the pelvis
* Prior history of chemotherapy for rectal cancer
* Active connective tissue disease such as scleroderma or Crohn's disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-10-26 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amol K Narang, M.D., Principal Investigator — Johns Hopkins Department of Radiation Oncology
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- High-dose Endorectal Brachytherapy (HDRBT): The investigational tool being evaluated is high-dose endorectal brachytherapy (HDRBT) which is an FDA approved method to administer endoluminal radiation for low rectal cancer.
  Daily dose of 6.5 Gy over four consecutive days
Period: Overall Study
Arm/Group | High-dose Endorectal Brachytherapy (HDRBT)
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- HDRBT: Radiation: High-dose endorectal brachytherapy The investigational tool being evaluated is high-dose endorectal brachytherapy (HDRBT) which is an FDA approved method to administer endoluminal radiation for low rectal cancer.
  High-dose endorectal brachytherapy: The investigational tool being evaluated is high-dose endorectal brachytherapy (HDRBT) which is an FDA approved method to administer endoluminal radiation for low rectal cancer.
Arm/Group | HDRBT
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pathologic Complete Response
Description: Those participants whose surgical pathology indicated that they had a complete response measured by RECIST.
  Per Response Evaluation Criteria In Solid Tumors (RECISTv1.0). Complete response (CR) indicating no tumors, a partial (PR) response indicating at least a 30% decrease in tumor diameter (PR), progressive disease (PD) indicating 20% or greater increase in tumor diameter, and stable disease (SD) indicating that the tumor did not shrink significantly to be considered a partial response and did not grow significantly enough to be considered progressive disease.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HDRBT (High Dose Rectal Brachytherapy)
Number analyzed (Participants) | 16
Participants | 5

2. Secondary Outcome: Number of Participants With Clinical Response of High-Dose-Rate Endorectal Brachytherapy (HDRBT) Brachytherapy
Description: Radiographic measurements of pelvic MRI and fluorodeoxyglucose (FDG) positron emission tomography (PET)/CT imaging will be used to classify patients as responders or non-responders to HDRBT using standard RECIST criteria.
  Response Evaluation Criteria In Solid Tumors (RECISTv1.0) is defined as follows: Complete response (CR) indicating no tumors, a partial (PR) response indicating at least a 30% decrease in tumor diameter (PR), progressive disease (PD) indicating 20% or greater increase in tumor diameter, and stable disease (SD) indicating that the tumor did not shrink significantly to be considered a partial response and did not grow significantly enough to be considered progressive disease.
Time Frame: 3 to 6 weeks post-treatment
Population: One patient had to go into surgery and it was not possible to do the imaging necessary for this assessment.
Measure: Count of Participants; unit: Participants
Groups:
- HDRBT: The investigational tool being evaluated is high-dose endorectal brachytherapy (HDRBT) which is an FDA approved method to administer endoluminal radiation for low rectal cancer.
  Daily dose of 6.5 Gy over four consecutive days
Arm/Group | HDRBT
Number analyzed (Participants) | 15
Participants
  Complete Response | 1
  Partial response | 13
  Progressive disease | 0
  Stable disease | 1

3. Secondary Outcome: Patient-reported Quality of Life (QOL) as Assessed by the EORTC QLQ-C30 Scores
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 form is a self-assessment completed by patients which examines current symptoms and functionality. Total score ranges from 0 to 100, a higher score represents a higher ("better") quality of life.
Time Frame: Pre-HDRBT, during HDRBT, post HDRBT week 1, week 2, weeks 3-6, 3-6 weeks post-op, every 4 months for 2 years and every 6 months for years 3 and 4
Population: Not all participants could be assessed at all the time points therefore data was not collected for some participants at some points as shown by participants for those time points being less than 16.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HDRBT
Number analyzed (Participants) | 16
score on a scale
  Pre-HDRBT | 47.5 (8.53)
  During HDRBT: number analyzed (Participants) | 10
  During HDRBT | 50 (12.45)
  1 week Post-HDRBT Treatment: number analyzed (Participants) | 13
  1 week Post-HDRBT Treatment | 52.23 (7.2)
  2 Weeks Post-HDRBT Treatment: number analyzed (Participants) | 3
  2 Weeks Post-HDRBT Treatment | 64.33 (10.69)
  3-6 weeks Post-HDRBT Treatment | 62.03 (13.09)
  3-6 weeks post-op: number analyzed (Participants) | 15
  3-6 weeks post-op | 59.27 (8.9)
  4 Months post-op: number analyzed (Participants) | 5
  4 Months post-op | 60.4 (13.11)
  8 Months post-op: number analyzed (Participants) | 5
  8 Months post-op | 53 (8.28)
  12 Months post-op: number analyzed (Participants) | 10
  12 Months post-op | 54 (9.48)
  16 Months post-op: number analyzed (Participants) | 9
  16 Months post-op | 49.89 (12.54)
  20 Months post-op: number analyzed (Participants) | 9
  20 Months post-op | 52.11 (6.27)
  24 Months post-op: number analyzed (Participants) | 10
  24 Months post-op | 56.5 (15.96)
  30 Months post-op: number analyzed (Participants) | 7
  30 Months post-op | 54.29 (13)
  36 Months post-op: number analyzed (Participants) | 8
  36 Months post-op | 56.5 (10.3)
  42 Months post-op: number analyzed (Participants) | 4
  42 Months post-op | 59.5 (7.23)
  48 Months post-op: number analyzed (Participants) | 4
  48 Months post-op | 53.75 (13.45)

4. Secondary Outcome: Patient-reported Quality of Life as Assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-CR38) Scores
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire QLQ-CR38 form is a self-assessment completed by patients and examine current symptoms and functionality. Each item is scored from 1 to 4. Total score range is from 38-152. A higher score represents better quality of life.
Time Frame: Pre-HDRBT, during HDRBT, post HDRBT week 1, week 2, weeks 3-6, 3-6 week post-op, every 4 months for 2 years and every 6 months for years 3 and 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HDRBT
Number analyzed (Participants) | 16
score on a scale
  Pre-HDRBT | 40.63 (7.37)
  During HDRBT: number analyzed (Participants) | 10
  During HDRBT | 36.8 (8.77)
  1 week Post-HDRBT Treatment: number analyzed (Participants) | 13
  1 week Post-HDRBT Treatment | 42.08 (11.24)
  2 Weeks Post-HDRBT Treatment: number analyzed (Participants) | 3
  2 Weeks Post-HDRBT Treatment | 42 (8.19)
  weeks 3-6 Post-HDRBT Treatment | 48.72 (17.62)
  3-6 weeks post-op: number analyzed (Participants) | 15
  3-6 weeks post-op | 47.8 (12.14)
  4 Months post-op: number analyzed (Participants) | 5
  4 Months post-op | 45.6 (4.34)
  8 Months post-op: number analyzed (Participants) | 5
  8 Months post-op | 50 (7.78)
  12 Months post-op: number analyzed (Participants) | 10
  12 Months post-op | 43.6 (11.53)
  16 Months post-op: number analyzed (Participants) | 9
  16 Months post-op | 47.67 (5.12)
  20 Months post-op: number analyzed (Participants) | 9
  20 Months post-op | 45 (6.54)
  24 Months post-op: number analyzed (Participants) | 10
  24 Months post-op | 47.3 (9.74)
  30 Months post-op: number analyzed (Participants) | 7
  30 Months post-op | 38.86 (20.76)
  36 Months post-op: number analyzed (Participants) | 8
  36 Months post-op | 49.75 (10.47)
  42 Months post-op: number analyzed (Participants) | 4
  42 Months post-op | 46 (2.16)
  48 Months post-op: number analyzed (Participants) | 4
  48 Months post-op | 38.75 (3.4)

5. Secondary Outcome: Patient-reported Quality of Life as Assessed by the European Organisation for Research and Treatment of Cancer, Quality of Life Questionnaire (EORTC QLQ-CR29) Scores
Description: The European Organisation for Research and Treatment of Cancer, Quality of Life Questionnaire (EORTC QLQ-CR29) form is a self-assessment completed by patients and examine current symptoms and functionality. Each item is scored from 1 to 4. Total score ranges from 29 - 116. A higher score represents better quality of life.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HDRBT
Number analyzed (Participants) | 16
score on a scale
  Pre-HDRBT | 34.56 (6.03)
  During HDRBT: number analyzed (Participants) | 10
  During HDRBT | 32.3 (5.27)
  1 week Post-HDRBT Treatment: number analyzed (Participants) | 13
  1 week Post-HDRBT Treatment | 37.46 (9.91)
  2 Weeks Post-HDRBT Treatment: number analyzed (Participants) | 3
  2 Weeks Post-HDRBT Treatment | 34 (11.53)
  3-6 weeks Post-HDRBT Treatment | 41.78 (14.62)
  3-6 weeks post-op: number analyzed (Participants) | 15
  3-6 weeks post-op | 42.6 (10.47)
  4 Months post-op: number analyzed (Participants) | 5
  4 Months post-op | 42.2 (3.96)
  8 Months post-op: number analyzed (Participants) | 5
  8 Months post-op | 43 (6.82)
  12 Months post-op: number analyzed (Participants) | 10
  12 Months post-op | 42 (6.78)
  16 Months post-op: number analyzed (Participants) | 9
  16 Months post-op | 41.22 (5.36)
  20 Months post-op: number analyzed (Participants) | 9
  20 Months post-op | 35.56 (6.78)
  24 Months post-op: number analyzed (Participants) | 10
  24 Months post-op | 40.2 (11.56)
  30 Months post-op: number analyzed (Participants) | 7
  30 Months post-op | 39.71 (12.72)
  36 Months post-op: number analyzed (Participants) | 8
  36 Months post-op | 43.5 (6.95)
  42 Months post-op: number analyzed (Participants) | 4
  42 Months post-op | 38.5 (6.56)
  48 Months post-op: number analyzed (Participants) | 4
  48 Months post-op | 30.75 (8.18)

6. Secondary Outcome: Number of Participants With Acute Gastrointestinal Toxicity Associated With High-Dose-Rate Endorectal Brachytherapy (HDRBT) as Assessed by CTCAE v4.0
Description: Acute gastrointestinal toxicity will be assessed using the Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.0). CTCAE v4.0 ratings of 3 or 4 (seriousness of 17%) adverse events will be assessed and reported.
Time Frame: 3-6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HDRBT (High Dose Rectal Brachytherapy)
Number analyzed (Participants) | 16
Participants
  Grade 3 pain | 2
  Grade 3 Proctitis | 1

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- High-Dose-Rate Endorectal Brachytherapy (HDRBT): The investigational tool being evaluated is high-dose endorectal brachytherapy (HDRBT) which is an FDA approved method to administer endoluminal radiation for low rectal cancer.
  Daily dose of 6.5 Gy over four consecutive days
Arm/Group | High-Dose-Rate Endorectal Brachytherapy (HDRBT)
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 3/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Dose-Rate Endorectal Brachytherapy (HDRBT) (N=16)
Pain (General disorders) | 2 (2)
Proctitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High-Dose-Rate Endorectal Brachytherapy (HDRBT) (N=16)
Pain (General disorders) | 16
Fatigue (General disorders) | 16
Anemia (Blood and lymphatic system disorders) | 16
Hyperglycemia (Metabolism and nutrition disorders) | 16
Constipation (Gastrointestinal disorders) | 13
Proctitis (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 10
Fecal Incontinence (Gastrointestinal disorders) | 10
GI - hemorrhage (Gastrointestinal disorders) | 10
Hemorrhoids (Gastrointestinal disorders) | 10
Rectal pain (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 9
WBC count decreased (Blood and lymphatic system disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 8
Lymphocyte count decreased (Blood and lymphatic system disorders) | 8
ALT increase (Metabolism and nutrition disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 6
Nocturia (Renal and urinary disorders) | 6
Urinary Frequency/urgency (Renal and urinary disorders) | 6
Dysuria (Renal and urinary disorders) | 5
Erectile dysfunction (General disorders) | 4
Neutrophil count decreased (Blood and lymphatic system disorders) | 4
Platelet count deceased (Blood and lymphatic system disorders) | 4
Urinary incontinence (Renal and urinary disorders) | 4
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 3
Aspartate Amino Transferase increased (Metabolism and nutrition disorders) | 3
AST increased (Metabolism and nutrition disorders) | 3
Hyponatremia (Blood and lymphatic system disorders) | 3
Urinary retention (Renal and urinary disorders) | 3
Alanine Amino Transferase Increased (Metabolism and nutrition disorders) | 2
Blood bilirubin increased (Blood and lymphatic system disorders) | 2
Incontinence (Renal and urinary disorders) | 2
Rectal Obstruction (Gastrointestinal disorders) | 2
Rectal stenosis (Gastrointestinal disorders) | 2
Vaginal dryness (Reproductive system and breast disorders) | 2
Vomiting (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes